CLINICAL TRIAL: NCT02365974
Title: Effects of Transcutaneous Electrical Nerve Stimulation (TENS) on Arterial Stiffness and Blood Pressure in Resistant Hypertensive Individuals
Brief Title: Transcutaneous Electrical Nerve Stimulation (TENS) on Arterial Stiffness and Blood Pressure
Acronym: TENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hospital de Base (Other)
Responsible Party: Principal Investigator, JOSE FERNANDO VILELA-MARTIN, Coordinator of Hypertension Clinic, Hospital de Base
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: RH-07606212500005415
Record Dates: First submitted 2015-02-08; First posted 2015-02-19 (Estimated); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: Hypertension; Vascular Stiffness; Autonomic Nervous System Diseases
Keywords: arterial stiffness; resistant hypertension; sympathetic system; blood pressure; transcutaneous electrical nerve stimulation
MeSH Terms: conditions — Hypertension; Autonomic Nervous System Diseases | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous Electrical Stimulation (Active Comparator): TENS will be applied in the cervicothoracic ganglion region located between the C7 and T4 vertebral processes for 40 minutes three times weekly for a total of four weeks. The intensity in milliamps (mA) will be adjusted depending on the sensitivity of each individual patient. The arrangement thereof will be parallel on each side of the C7 (channel 1) and T4 (channel 2) vertebral spinous processes.
  Interventions: Device: Transcutaneous Electrical Stimulation
- No Transcutaneous Electrical Stimulation (Sham Comparator): The sham group will be submitted to the procedure to fit the stimulation equipment without be submitted to stimulation.
  Interventions: Device: No Transcutaneous Electrical Stimulation

INTERVENTIONS:
Device: Transcutaneous Electrical Stimulation — TENS will be applied in the cervicothoracic ganglion region located between the C7 and T4 vertebral processes for 40 minutes three times weekly for a total of four weeks. The intensity in milliamps will be adjusted depending on the sensitivity of each individual patient.
  Arms: Transcutaneous Electrical Stimulation
Device: No Transcutaneous Electrical Stimulation — The sham group will be submitted to the procedure to fit the stimulation equipment. without be submitted to stimulation.
  Arms: No Transcutaneous Electrical Stimulation

SUMMARY:
Uncontrolled blood pressure represents the main factor in the development of target organ lesions and, consequently, cardiovascular events, which are the leading cause of morbidity and mortality worldwide. In most cases resistant hypertension is preceded by target organ lesions, and is strongly influenced by risk factors or associated diseases. To control this disease requires an adequate and intense therapeutic approach that includes lifestyle changes and the use of several antihypertensive drugs. However, the results are not always satisfactory despite intensive treatment. Of the different pathophysiological mechanisms involved in the pathogenesis of resistant hypertension (RH), two, sympathetic overstimulation and therapies that block the sympathetic system, have been widely studied. But, these approaches are invasive and expensive. Another possible approach is by transcutaneous electrical nerve stimulation (TENS), a non-invasive method that modulates activity by inhibiting primary afferent pathways using low-frequency transcutaneous electrical stimulation. Some studies have shown that TENS reduces blood pressure in patients with hypertension. The current study will evaluate the effect of applying TENS in the cervicothoracic region of subjects with resistant hypertension, seeking to develop a new low cost and readily available therapy to treat this group of hypertensive individuals.

DETAILED DESCRIPTION:
Patients will be divided into two groups: treatment and control (sham group). The sham group will be submitted to the procedure to fit the stimulation equipment. However, these patients will not be submitted to stimulation. Both groups will undergo a physical examination at the start and end of the study period to determine anthropometric variables. The BMI, defined as the weight (kg) divided by the patient's height squared (m2), will be calculated. The height will be determined in centimeters using a measuring tape with the individual barefoot. Individuals with BMI <25 kg/m² will be classified as normal, overweight as a BMI between 25 and 30 kg/m², and obese as a BMI ≥30 kg/m². The waist circumference will be measured using a measuring tape at half the distance between the iliac crest and the lower costal margin. Patients will undergo the following tests before and after the end of the four-week study period: 24-hour ambulatory blood pressure monitoring (ABPM), 24-hour dynamic electrocardiography, continuous measurement of beat-to-beat BP, endothelial function measurement and radial artery applanation tonometry (AT).

Biochemical tests will be performed at two time points, before and after the four-week study period and include blood sugar, total cholesterol (TC), high-density lipoprotein cholesterol (HDL-C), triglycerides (TG), creatinine, potassium, uric acid, and plasma insulin levels. Blood sugar, TC, HDL-C and TG levels will be determined by colorimetry after fasting for 12 hours using a dimension device with the Dade Behring reagent. Diagnosis of diabetes mellitus (DM) will be established by patient history, the use of hypoglycemic drugs and measurement of the serum glucose. The LDL-C fraction will be calculated using the formula LDL-C = TC - HDL-C - TG / 5 (for TG <400 mg/dL). Additionally, the electrochemiluminescence method will be used to measure plasma insulin (immunoassay for the in vitro quantitative determination of human insulin in serum and plasma using the Elecsys 1010/2010 immunoassay and E170 modular analytics analyzers by Roche). The homeostasis model assessment of insulin resistance (HOMA-IR) index will be applied after obtaining blood sugar and insulin levels in order to determine insulin resistance and the functional capability of the pancreatic beta cells. Insulin resistance will be characterized when this ratio exceeds 2.71. The HOMA-IR index is calculated using the following formula:

HOMA-IR: Fasting insulin (McU/mL) x fasting glucose (mmol/L*) 22.5

In order to convert the glucose concentration to mmol/L it is necessary to multiply the value in mg/dL by 0.0555. Measurement of serum creatinine will be performed by a standardized enzyme-kinetic biochemical test and will be considered high when serum creatinine >1.4 mg/dL. Urinary sodium and potassium levels (mEq/L) will be evaluated by flame photometry. Urinary sodium excretion will be calculated by multiplying the urinary sodium and potassium concentrations in mEq/L by the 24-hour urine volume. The 24-hour urine volume and urinary creatinine concentrations will be assessed to calculate creatinine clearance adjusted for body surface.

Specific biochemical tests will be considered: serum aldosterone (AS), plasma renin activity (PRA), high-sensitivity C-reactive protein (hsCRP), metalloproteinase 9 (MMP-9), tissue inhibitor of metalloproteinases (TIMP-1 and TIMP-2), nitrites and nitrates, interleukin-1, 6, 8, 10 and 18 (IL-1, IL-6, IL-8, IL-10 and IL-18), tumor necrosis factor (TNF-α), thromboxane B2 (TXB2), fibrinogen, intercellular adhesion molecule (ICAM-1), plasminogen activator inhibitor (PAI-1), angiotensin converting enzyme (ACE) and angiotensin II (Ang II).

ELIGIBILITY:
Inclusion Criteria:

* RH patients taking at least three antihypertensive drugs at full doses, one of which is preferably a thiazide diuretic; Age between 40 and 70 years.

Exclusion Criteria:

* Use of a cardiac pacemaker
* Cardiac electrical conduction abnormalities evidenced by ECG or stress test (ergometry)
* Dermatological abnormalities at the site of the application of TENS
* Uncontrolled diabetes patients using oral hypoglycemic agents or insulin with glycated Hb ≥ 7.5%
* Secondary Hypertension
* Patients who do not adhere to the lifestyle changes recommended by their physician such as low-sodium diet and weight loss
* Moderate to severe cervical-thoracic scoliosis
* Obesity with body mass index (BMI) ≥35 kg/m2

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2021-06-01 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in peripheral blood pressure of individuals with resistant hypertension after transcutaneous electrical nervous stimulation. | 30 days

SECONDARY OUTCOMES:
Change from baseline in central blood pressure of individuals with resistant hypertension after transcutaneous electrical nervous stimulation. | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: José F Vilela-Martin, MD PhD, Principal Investigator — Fundação Faculdade Regional de Medicina de São José do Rio Preto

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] da Silva ML, Chiappa GR, da Silva VM, Neves LM, de Lima AC, Tomasi FP, Junior LT, Vilela-Martin JF, Bottaro M, Junior GC. Effect of transcutaneous electrical nerve stimulation on peripheral to central blood pressure ratio in healthy subjects. Clin Physiol Funct Imaging. 2016 Jul;36(4):293-7. doi: 10.1111/cpf.12227. Epub 2015 Jan 30. PMID 25640037
- [Background] Cipriano G Jr, Neder JA, Umpierre D, Arena R, Vieira PJ, Chiappa AM, Ribeiro JP, Chiappa GR. Sympathetic ganglion transcutaneous electrical nerve stimulation after coronary artery bypass graft surgery improves femoral blood flow and exercise tolerance. J Appl Physiol (1985). 2014 Sep 15;117(6):633-8. doi: 10.1152/japplphysiol.00993.2013. Epub 2014 Aug 7. PMID 25103974
- [Derived] Vilela-Martin JF, Giollo-Junior LT, Chiappa GR, Cipriano-Junior G, Vieira PJ, dos Santos Ricardi F, Paz-Landim MI, de Andrade DO, Cestario Edo E, Cosenso-Martin LN, Yugar-Toledo JC, Cipullo JP. Effects of transcutaneous electrical nerve stimulation (TENS) on arterial stiffness and blood pressure in resistant hypertensive individuals: study protocol for a randomized controlled trial. Trials. 2016 Mar 29;17:168. doi: 10.1186/s13063-016-1302-8. PMID 27026087